CLINICAL TRIAL: NCT06200558
Title: ARON-3 Study: International Multicentric Retrospective Study to Collect Global Experiences in the Treatment of Patients With Metastatic PCa
Status: Recruiting | Type: Observational
Sponsor: Hospital of Macerata (Other)
Responsible Party: Principal Investigator, Matteo Santoni, Medical Doctor, Principal Investigator, Hospital of Macerata
Other Study IDs: ARON-3
Record Dates: First submitted 2023-12-03; First posted 2024-01-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: mCSPC; Lutetium-177 PSMA; PARP inhibitors; ADT; ARSI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- For ARON-3S: Patients with metachronous or de novo metastatic hormone/castration-sensitive PCa: Patients with metachronous or de novo metastatic hormone/castration-sensitive PCa treated with ADT+ARSI or ADT+ARSI+docetaxel
- For ARON-3Lu: Patients receiving Lutetium-177 PSMA for castration resistant PC (CRPC)
- For ARON-3GEN: Patients treated with PARP inhibitors (alone or plus ARSI) for CRPC

SUMMARY:
Study wants to explore real-world data in three distinct settings

* Patients with metachronous or de novo mCSPC treated with ADT+ARSI or ADT+ARSI+docetaxel _ARON-3S
* Patients receiving Lutetium-177 PSMA for mCRPC _ ARON-3Lu
* Patients treated with PARP inhibitors (alone or combined with ARSI) for CRPC _ ARON-3GEN

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18y
* Cytological or Histologically confirmed diagnosis of PC
* Histologically or radiologically confirmed diagnosis of metastatic disease and

For ARON-3S

▪ Treatment with ADT + Apalutamide or ADT + enzalutamide or ADT + Abiraterone or ADT + Abiraterone + Docetaxel or ADT + Darolutamide + Docetaxel (patients treated with previous docetaxel - CHAARTED - resulted eligible)

For ARON-3Lu

▪ Treatment with Luthetium-177-PSMA therapy for castration resistant PC

For ARON-3GEN

* HRD POSITIVE STATUS
* Treatment with PARP inhibitors for castration resistant PC. Treatment included: olaparib (as 1st, 2nd or 3rd line therapy), olaparib + abiraterone (as 1st line therapy) or niraparib + abiraterone (as 1st line therapy) or talazoparib + enzalutamide

Exclusion Criteria:

* Patients without histologically confirmed diagnosis of PC
* Patients without histologically or radiologically confirmed metastatic disease and

For ARON-3S

▪ Patients treated with doublets or triplets not included in the list reported in the Inclusion Criteria Section

For ARON-3Lu

▪ Patients treated with Luthetium-177-PSMA therapy for hormone/castration sensitive PC

For ARON-3GEN

* HRD NEGATIVE STATUS
* Patients treated with PARP inhibitors alone or in combination regimens not included in the ARON-3GEN study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment of patients with metastatic PCa. In the ARON-3 Study the investigators focused on three different settings:
  * ARON-3S: Patients with metachronous or de novo metastatic hormone/castration-sensitive PCa treated with ADT + ARSI or ADT + ARSI + docetaxel
  * ARON-3Lu: Patients receiving Lutetium-177 PSMA for castration resistant PC (CRPC)
  * ARON-3GEN: Patients treated with PARP inhibitors (alone or plus ARSI) for CRPC
Sampling Method: Non-Probability Sample
Enrollment: 534 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) of patients with hormone/castration-sensitive PC treated with ADT + ARSI or ADT + ARSI + docetaxel | January 31h, 2024- May 31th, 2024
Progression-Free Survival of patients with hormone/castration-sensitive PC treated with ADT + ARSI or ADT + ARSI + docetaxel | January 31h, 2024- May 31th, 2024
Overall Response Rate of patients with hormone/castration-sensitive PC treated with ADT + ARSI or ADT + ARSI + docetaxel | January 31h, 2024- May 31th, 2024
Overall Survival (OS) of patients with castration resistant PC treated with Luthetium-177-PSMA therapy | January 31h, 2024- May 31th, 2024
Progression-Free Survival (PFS) of patients with castration resistant PC treated with Luthetium-177-PSMA therapy | January 31h, 2024- May 31th, 2024
Overall Response Rate (ORR) of patients with castration resistant PC treated with Luthetium-177-PSMA therapy | January 31h, 2024- May 31th, 2024
Overall Survival (OS) of patients with castration resistant PC treated with PARP inhibitors alone or in combined regimens | January 31h, 2024- May 31th, 2024
Progression-Free Survival (PFS) of patients with castration resistant PC treated with PARP inhibitors alone or in combined regimens | January 31h, 2024- May 31th, 2024
Overall Response Rate (ORR) of patients with castration resistant PC treated with PARP inhibitors alone or in combined regimens | January 31h, 2024- May 31th, 2024

SECONDARY OUTCOMES:
Time to progression of patients with different metastatic sites treated by the distinct combinations | January 31h, 2024- May 31th, 2024
  Statistical analysis of data obtained by medical charts related to disease metastatic sites, treatment performed and period of time from the start of treatment until the radiological progression disease
prognostic role of lifestyle and concomitant medications | January 31h, 2024- May 31th, 2024
  Statistical analysis of data obtained by medical charts related to lifestyle and concomitant medications

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale di Macerata, Macerata, Macerata, Italy